CLINICAL TRIAL: NCT00464581
Title: A Single-center Phase 2 Trial of Intravitreous Injections of Lucentis (Ranibizumab) in Subjects With Cystoid Macular Edema Secondary to Non-ischemic Retinopathy
Brief Title: Lucentis for Treatment of Macular Edema
Acronym: FVF4153s
Status: Completed | Type: Observational
Sponsor: Retina Institute of Hawaii (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Debbie Shimabukuro, Study Coordinator, Retina Institute of Hawaii
Other Study IDs: FVF-4153s
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Cystoid Macular Edema
Keywords: non-ischemic retinopathy
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cystoid macular edema (CME) is the most common cause of suboptimal post-operative visual acuity in uncomplicated cataract extractions. Over two million cataract extractions are performed each year, with a reported incidence ranging from 1.5 to 6.9%, resulting in an estimated 20,000-130,000 new cases of CME annually. Clinical CME historically was associated with visual acuity of 20/40 or worse with fluorescein angiographic evidence of macular edema in a classic petaloid pattern. Angiographic CME physiologically signals an inflammatory process causing distortion of the outer plexiform layer, which if not resolved quickly could result in non-repairable visual loss. Topical, periocular, or intravitreal corticosteroids, despite their associated side effects, are the mainstay for pharmacologic treatment for patients with CME. Their efficacy has never been demonstrated in a randomized, controlled and blinded study.

This is an open-label, Phase II study of intravitreally administered ranibizumab in subjects with cystoid macular edema secondary to non-ischemic retinopathy, as seen following cataract surgery with intraocular lens implantation.

DETAILED DESCRIPTION:
Vascular endothelial growth factor (VEGF) is known to be induced by hypoxia and has been implicated in the development of iris and retinal vascularization. VEGF, however, is also known to be a potent mediator of vascular permeability in other tissues and may perform this function in retina.

Immunohistochemical VEGF staining has been identified in patients with disorders such as aphakic and pseudophakic cystoid macular edema, ocular inflammatory disease and infection. VEGF was primarily localized within retinal neurons and within the retinal pigment epithelium in these cases. In addition or in association with its role of inducing neovascularization (Wet AMD and diabetic retinopathy, VEGF may contribute to the breakdown of the blood-retinal barrier in a variety of disorders.

Ranibizumab is a pan-VEGF A blocker that has been proven highly effective for the treatment of wet macular degeneration. The underlying pathophysiology of both cystoid macular edema and wet AMD is VEGF overproduction.

To date ranibizumab has been approved only for treating wet ARMD. In this study we will explore ranibizumab for the treatment of cystoid macular edema It is hypothesized that this population will show dramatic improvement as the initial cause of VEGF production can be isolated to the surgical procedure and due to the fact that the retinal pigment epithelium is healthier in this population as compared to the macular degeneration counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age < 90 years
* Cystoid macular edema, documented by FFA
* Best corrected visual acuity in the study eye between 85 and 20 ETDRS letters or between 20/30 and 20/800 in a Snellen chart.
* Women must be using two forms of effective contraception, be post¬menopausal for at least 12 months prior to trial entry, or surgically sterile; if of child-bearing potential, a urine pregnancy test must be performed within 7 days prior to the first injection with a negative result. If the test is positive, a serum test must be done to confirm. The two forms of effective contraception must be implemented during the trial and for at least 60 days following the last dose of test medication.

Exclusion Criteria:

* Significant media opacities, which might interfere with visual acuity.
* Any ocular or periocular infection in the past 4 weeks.
* Presence of pigment epithelial tears or rips.
* Any of the following underlying diseases including:

  * Diabetic retinopathy.
  * History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 16.6), clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within 6 months, ventricular tachyarrhythmias requiring ongoing treatment.
  * History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
  * History or evidence of clinically significant impaired renal or hepatic function
  * Stroke (within 12 months of trial entry).
  * Any major surgical procedure within one month of trial entry.
* Previous therapeutic radiation in the region of the study eye.
* Any treatment with an investigational agent in the past 30 days for any condition.
* Known serious allergies to the fluorescein dye used in angiography or to the components of ranibizumab formulation.

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Macular Edema
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ranibizumab in patients with CME secondary to non-ischemic retinopathy | 2 years

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart, at each month of months 0-12. | 2 years
Proportion of subjects who remained at baseline VA or gained >0 lines of vision from baseline to week 24 and 52. | 2 years
Mean change in central retinal thickness on OCT 3 from Baseline to week 24 and 52. | 2 years
Changes observed on the Fluoreosceiien Angiographs from baseline to week 24 and 52. | 2 years
Mean number of ranibizumab injections required. | 2 years
Nidek MPI measurements taken at baseline, week 24, and week 52 | 2 years
Proportion of subjects who demonstrate complete resolution of macular edema as seen on OCT testing from baseline to week 52 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Bennett, MD, Principal Investigator — Retina Institute of Hawaii
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States